CLINICAL TRIAL: NCT05153005
Title: Comprehensive Diagnosis and Treatment Strategy for Opportunistic Fungal Infections in AIDS Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou 8th People's Hospital (Other)
Responsible Party: Principal Investigator, Linghua LI, Chief physician, Guangzhou 8th People's Hospital
Other Study IDs: 202034167
Record Dates: First submitted 2021-11-15; First posted 2021-12-10 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Opportunistic Fungal Infections
Keywords: Talaromycosis; Pneumocystis pneumonia; Cryptococcus Infection
MeSH Terms: conditions — talaromycosis; Pneumonia, Pneumocystis; Cryptococcosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Talaromycosis: Participants: AIDS patients complicated with Talaromycosis. Intervention(s): To use the specific antigen of taloromyces marneffei which is mannose protein (Mp1p), (1,3)- β- D-glucan (G antigen) and qPCR, dd-PCR and mass spectrometry identification in the diagnosis and efficacy evaluation of AIDS patients complicated with Talaromycosis.
  Interventions: Other: examination methods
- Pneumocystis pneumonia: Participants: AIDS patients complicated with Pneumocystis pneumonia Intervention(s)：To use (1,3)- β- D-glucan (G antigen) , qPCR, dd-PCR and mass spectrometry identification, to explore the methods of screening and early diagnosis strategies.
  Interventions: Other: examination methods
- Cryptococcus: Participants: AIDS patients complicated with Cryptococcus Intervention(s)：To use (1,3)- β- D-glucan (G antigen) and Cryptococcus capsular antigen(CrAg) serological detection, qPCR, DD PCR and mass spectrometry identification, to explore the methods of screening and early diagnosis strategies of disease.
  Interventions: Other: examination methods

INTERVENTIONS:
Other: examination methods — Some advanced methods: mannose protein (Mp1p), (1,3)- β- D-glucan (G antigen) and Cryptococcus capsular antigen (CrAg) serological detection, qPCR, dd- PCR and mass spectrometry identification, QFC.

SUMMARY:
Opportunistic fungal infection is the most common opportunistic infection in AIDS patients, with the high mortality and recurrence rate due to the lack of standardized comprehensive diagnosis and treatment strategy. This project aims to combine traditional detection and observation indicators with molecular biology, serology and mass spectrometry identification technology to develop early screening and diagnostic strategies for opportunistic fungal infections in AIDS patients, explore scientific evaluation methods for anti-fungal efficacy and formulate comprehensive strategies for reducing the mortality and recurrence rate.

DETAILED DESCRIPTION:
The research involves AIDS patients complicated with talaromycosis, PCP and cryptococcosis in the study.

The main contents:

1. To explore early screening and diagnostic strategies. To advance the application of taloromyces marneffeispecific mannose protein (Mp1p), (1,3)- β- D-glucan (G antigen) and Cryptococcus capsular antigen (CrAg) serological detection, qPCR, dd- PCR and mass spectrometry identification In clinical practice.
2. To develop scientific evaluation strategy of anti-fungal treatment effect. On the basis of routine clinical, laboratory, imaging indexes and QFC, qPCR, dd-PCR and serological quantitative detection methods were combined to explore strategies for evaluating anti-fungal efficacy. 3 .To determine the termination timing of secondary prevention To explore the scientific timing to terminate secondary prevention after ART, Combing CD4 + T cell count with plasma HIV RNA, HIV DNA of peripheral blood mononuclear cells (PBMC), CD4 + / CD8+ ratio and chronic immune activation index

ELIGIBILITY:
Inclusion Criteria:

1. Age (16-70 years), male and female;
2. HIV-1 infected;
3. hospitalized patients with the signs or symptoms inferred to infection;
4. Initial CD4 cell count less than 200 cells/ul; HIV-1 RNA viral load was unlimited;
5. State Informed Consent for Free Treatment has been signed;
6. Good compliance and signing Informed Consent

Exclusion Criteria:

1. have been treated regularly in other hospitals or have been clearly diagnosed before admission;
2. Researchers decide if patients could/not complete the scheduled follow-up (factors to consider such as weak, poor compliance, etc.);
3. Pregnancy during the study period;
4. Hospital stay less than 7 days.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population for screening of important opportunistic fungal infections: About 2000 AIDS patients, with CD4 + < 200 cells /μ, regardless of whether they received ART or not.
  Population for efficacy evaluation: about 420 patients with AIDS complicated with Talaromycosis, PCP or cryptococcosis.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of patients who achieved etiological diagnosis of opportunistic fungal infection | 2 weeks
  The probability of etiological diagnosis achieved by new diagnostic techniques after admission
Number of hospitalized patients who achieved clinical remission or cure | 6 months
  The improvement of treatment efficiency for treating with 3 main opportunistic fungal infections in AIDS patients when applying with new diagnostic techniques

CONTACTS AND LOCATIONS:
Overall Officials: Ruosu Ying, PhD, Study Director — Guangzhou Eighth People's Hospital, Guangzhou Medical University
Locations (1):
- Guangzhou Eighth People's Hospital, Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] IeDEA and ART Cohort Collaborations; Avila D, Althoff KN, Mugglin C, Wools-Kaloustian K, Koller M, Dabis F, Nash D, Gsponer T, Sungkanuparph S, McGowan C, May M, Cooper D, Chimbetete C, Wolff M, Collier A, McManus H, Davies MA, Costagliola D, Crabtree-Ramirez B, Chaiwarith R, Cescon A, Cornell M, Diero L, Phanuphak P, Sawadogo A, Ehmer J, Eholie SP, Li PC, Fox MP, Gandhi NR, Gonzalez E, Lee CK, Hoffmann CJ, Kambugu A, Keiser O, Ditangco R, Prozesky H, Lampe F, Kumarasamy N, Kitahata M, Lugina E, Lyamuya R, Vonthanak S, Fink V, d'Arminio Monforte A, Luz PM, Chen YM, Minga A, Casabona J, Mwango A, Choi JY, Newell ML, Bukusi EA, Ngonyani K, Merati TP, Otieno J, Bosco MB, Phiri S, Ng OT, Anastos K, Rockstroh J, Santos I, Oka S, Somi G, Stephan C, Teira R, Wabwire D, Wandeler G, Boulle A, Reiss P, Wood R, Chi BH, Williams C, Sterne JA, Egger M. Immunodeficiency at the start of combination antiretroviral therapy in low-, middle-, and high-income countries. J Acquir Immune Defic Syndr. 2014 Jan 1;65(1):e8-16. doi: 10.1097/QAI.0b013e3182a39979. PMID 24419071
- [Background] Waldrop G, Doherty M, Vitoria M, Ford N. Stable patients and patients with advanced disease: consensus definitions to support sustained scale up of antiretroviral therapy. Trop Med Int Health. 2016 Sep;21(9):1124-30. doi: 10.1111/tmi.12746. Epub 2016 Jul 22. PMID 27371814
- [Background] Tanuma J, Lee KH, Haneuse S, Matsumoto S, Nguyen DT, Nguyen DT, Do CD, Pham TT, Nguyen KV, Oka S. Incidence of AIDS-Defining Opportunistic Infections and Mortality during Antiretroviral Therapy in a Cohort of Adult HIV-Infected Individuals in Hanoi, 2007-2014. PLoS One. 2016 Mar 3;11(3):e0150781. doi: 10.1371/journal.pone.0150781. eCollection 2016. PMID 26939050
- [Background] Luo B, Sun J, Cai R, Shen Y, Liu L, Wang J, Zhang R, Shen J, Lu H. Spectrum of Opportunistic Infections and Risk Factors for In-Hospital Mortality of Admitted AIDS Patients in Shanghai. Medicine (Baltimore). 2016 May;95(21):e3802. doi: 10.1097/MD.0000000000003802. PMID 27227959
- [Background] Limper AH, Adenis A, Le T, Harrison TS. Fungal infections in HIV/AIDS. Lancet Infect Dis. 2017 Nov;17(11):e334-e343. doi: 10.1016/S1473-3099(17)30303-1. Epub 2017 Jul 31. PMID 28774701
- [Background] Jarvis JN, Govender N, Chiller T, Park BJ, Longley N, Meintjes G, Bekker LG, Wood R, Lawn SD, Harrison TS. Cryptococcal antigen screening and preemptive therapy in patients initiating antiretroviral therapy in resource-limited settings: a proposed algorithm for clinical implementation. J Int Assoc Physicians AIDS Care (Chic). 2012 Nov-Dec;11(6):374-9. doi: 10.1177/1545109712459077. Epub 2012 Sep 26. PMID 23015379
- [Background] Beyene T, Zewde AG, Balcha A, Hirpo B, Yitbarik T, Gebissa T, Rajasingham R, Boulware DR. Inadequacy of High-Dose Fluconazole Monotherapy Among Cerebrospinal Fluid Cryptococcal Antigen (CrAg)-Positive Human Immunodeficiency Virus-Infected Persons in an Ethiopian CrAg Screening Program. Clin Infect Dis. 2017 Nov 29;65(12):2126-2129. doi: 10.1093/cid/cix613. PMID 29020172
- [Background] Kim YJ, Woo JH, Kim MJ, Park DW, Song JY, Kim SW, Choi JY, Kim JM, Han SH, Lee JS, Choi BY, Lee JS, Kim SS, Kee MK, Kang MW, Kim SI. Opportunistic diseases among HIV-infected patients: a multicenter-nationwide Korean HIV/AIDS cohort study, 2006 to 2013. Korean J Intern Med. 2016 Sep;31(5):953-60. doi: 10.3904/kjim.2014.322. Epub 2016 Apr 27. PMID 27117317
- [Background] Pruksaphon K, Intaramat A, Ratanabanangkoon K, Nosanchuk JD, Vanittanakom N, Youngchim S. Development and characterization of an immunochromatographic test for the rapid diagnosis of Talaromyces (Penicillium) marneffei. PLoS One. 2018 Apr 11;13(4):e0195596. doi: 10.1371/journal.pone.0195596. eCollection 2018. PMID 29641620
- [Background] Song Y, Ren Y, Wang X, Li R. Recent Advances in the Diagnosis of Pneumocystis Pneumonia. Med Mycol J. 2016;57(4):E111-E116. doi: 10.3314/mmj.16-00019. PMID 27904052